CLINICAL TRIAL: NCT00354796
Title: The Effect of Reduced Dose of Enoxaparin on the Laboratory and Clinical Outcomes of Treatment With Enoxaparin
Brief Title: The Effect of Reduced Dose of Enoxaparin on the Outcomes of Treatment With Enoxaparin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Mordechai Muszkat, Hadassah University Hospital
Other Study IDs: enoxap-HMO-CTIL
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Acute Coronary Syndrome; Venous Thromboembolism; Atrial Fibrillation; Hypercoagulability
Keywords: bleeding; anticoagulation; LMWH; Enoxaparin
MeSH Terms: conditions — Acute Coronary Syndrome; Venous Thromboembolism; Atrial Fibrillation; Thrombophilia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We hypothesize that reduced dose of enoxaparin in elderly patients will result in reduced proportion of patients with therapeutic anti Xa activity and reduced clinical efficacy.

DETAILED DESCRIPTION:
Patients treated with enoxaparin will be followed, sociodemographic , clinical and laboratory data will be collected. Clinical efficacy as well as adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* treatment with enoxaparin

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-07; Study Completion 2015-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Muszkat, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel